CLINICAL TRIAL: NCT05959018
Title: Efficacy & Health Economics of Antimicrobial-impregnated Central Venous Catheters (CVCs) Compared to Non-impregnated CVCs in Central Line-associated Bloodstream Infection Prevention in a Malaysia University Hospital Adult ICU
Brief Title: Efficacy & Cost Effectiveness of Antimicrobial-impregnated CVCs in CLABSI Prevention in a Malaysia Adult ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Teleflex (Industry)
Responsible Party: Principal Investigator, Tan Kai Ming, Principal Investigator/ Postgraduate Student, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UM-AMCVC-01
Record Dates: First submitted 2023-06-20; First posted 2023-07-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: CLABSI - Central Line Associated Bloodstream Infection
Keywords: Antimicrobial-impregnated Central Venous Catheters (CVCs); Central Line-associated Bloodstream Infection (CLABSI); Intensive Care Unit (ICU)

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Non-impregnated CVC - Arrow Three-Lumen Central Venous Catheter (Sham Comparator): Control group who receives non-impregnated CVC - Arrow Three-Lumen Central Venous Catheter
  Interventions: Device: Arrow Three-Lumen Central Venous Catheter
- Antimicrobial-impregnated CVC - Arrowg+ard Blue Plus® Three-Lumen Central Venous Catheter (Experimental): Group who receives antimicrobial-impregnated CVC - Arrowg+ard Blue Plus® Three-Lumen Central Venous Catheter
  Interventions: Device: Arrowg+ard Blue Plus® Three-Lumen Central Venous Catheter

INTERVENTIONS:
Device: Arrow Three-Lumen Central Venous Catheter — Participants in the Non-impregnated CVC arm will receive Arrow Three-Lumen Central Venous Catheter inserted by healthcare personnel for critical care use
  Arms: Non-impregnated CVC - Arrow Three-Lumen Central Venous Catheter
Device: Arrowg+ard Blue Plus® Three-Lumen Central Venous Catheter — Participants in the Antimicrobial-impregnated CVC arm will receive Arrowg+ard Blue Plus® Three-Lumen Central Venous Catheter inserted by healthcare personnel for critical care use
  Arms: Antimicrobial-impregnated CVC - Arrowg+ard Blue Plus® Three-Lumen Central Venous Catheter

SUMMARY:
Central venous catheters (CVCs) are indispensable in modern critical care. However, CVC usage is associated with complications, including central line-associated bloodstream infections (CLABSIs), which in turn, is translated to higher healthcare costs and mortality.

The use of antimicrobial-impregnated CVCs is one of the strategies to reduce CLABSI.

Nevertheless, its' efficacy and beneficial effects, particularly in terms of patients' outcome had not been homogeneously demonstrated across literature. Moreover, antimicrobial-impregnated CVCs are more expensive compared to conventional non-impregnated ones, and hence its cost-effectiveness remains doubtful. To date, no local studies have been conducted to evaluate the efficacy and economic impact of antimicrobial-impregnated CVCs and on patients' outcome.

The goal of this clinical trial is to determine the efficacy and cost-effectiveness of antimicrobial-impregnated CVCs in preventing (CLABSI) among critically ill patients in a Malaysia University Hospital Adult Intensive Care Unit.

The main questions it aims to answer are:

1. Is there any difference in CLABSI rates between patients using antimicrobial-impregnated CVCs and non-impregnated CVCs in Malaysia adult ICU?
2. Does the use of antimicrobial-impregnated CVCs in CLABSI prevention in Malaysia adult ICU affect patient length of stay when compared to non- impregnated CVCs?
3. Does the use of antimicrobial-impregnated CVCs in CLABSI prevention in the adult ICU setting affect healthcare costs when compared to non-impregnated CVCs?
4. How antimicrobial resistance features of the bacteria causing CLABSI may differ in patients using antimicrobial-impregnated CVCs compared to non-impregnated CVCs?

Patients who require a CVC for critical care in ICU will be recruited and randomly assigned to one of the two different groups to receive either a conventional non-impregnated CVC or an antimicrobial-impregnated CVC, which will be inserted and handled by medical practitioners. Participants will then be monitored for symptoms and signs of CLABSI, alongside length of ICU stay & healthcare costs. Researchers will compare CLABSI rates and other relevant parameters among the 2 groups to see if antimicrobial-impregnated CVCs are useful and cost-effective in CLABSI prevention.

DETAILED DESCRIPTION:
Central venous catheters (CVCs) are indispensable in modern critical care. The average central line utilisation ratios in the ICUs across 45 countries were reported at 0.525.

However, CVC usage is associated with complications, including central line-associated bloodstream infections (CLABSIs). The rate of CLABSI is reported at 4.45 per 1000 central line days in ICUs across 45 countries from 2013 - 2018. This in turn, is translated to higher healthcare costs and mortality.

Antimicrobial-impregnated CVCs are proposed to be able to reduce the incidence of CLABSI by inhibiting microorganism colonisation on CVCs. A meta-analysis published in 2018 concluded that antimicrobial-impregnated CVCs were significantly effective in reducing CLABSIs and catheter colonisations.

Nevertheless, its' efficacy and beneficial effects, particularly in terms of patients' outcome had not been homogeneously demonstrated across literature. Moreover, antimicrobial-impregnated CVCs are more expensive compared to conventional non-impregnated ones, and hence its' cost-effectiveness remains doubtful. To date, no local studies have been conducted to evaluate the efficacy and economic impact of antimicrobial-impregnated CVCs and on patients' outcome.

The goal of this clinical trial is to determine the efficacy and cost-effectiveness of antimicrobial-impregnated CVCs in preventing (CLABSI) among critically ill patients in a Malaysia University Hospital Adult Intensive Care Unit.

The main questions it aims to answer are:

1. Is there any difference in CLABSI rates between patients using antimicrobial-impregnated CVCs and non-impregnated CVCs in Malaysia adult ICU?
2. Does the use of antimicrobial-impregnated CVCs in CLABSI prevention in Malaysia adult ICU affect patient length of stay when compared to non-impregnated CVCs?
3. Does the use of antimicrobial-impregnated CVCs in CLABSI prevention in the adult ICU setting affect healthcare costs when compared to non-impregnated CVCs?
4. How antimicrobial resistance features of the bacteria causing CLABSI may differ in patients using antimicrobial-impregnated CVCs compared to non-impregnated CVCs?

The primary and secondary objectives of the study include the following:

- Primary objective: To compare the incidence of CLABSI rate in patients using antimicrobial-impregnated CVCs and non-impregnated CVCs in Malaysia adult ICU

- Secondary objectives:

1. To determine the length of stay of patients using antimicrobial-impregnated CVCs vs non-impregnated CVCs in Malaysia adult ICU
2. To undertake a cost-effectiveness analysis in prevention of CLABSI between patients using antimicrobial-impregnated CVCs and non-impregnated CVCs in Malaysia adult ICU
3. To compare the antimicrobial resistance features of the bacterial species that caused CLABSI between patients using antimicrobial-impregnated CVCs and that of non-impregnated CVCs in Malaysia adult ICU The study will be conducted in the adult Intensive Care Unit (ICU) of Universiti Malaya Medical Centre (UMMC), Malaysia, which is a mixed medical/surgical ICU, over a period of 1 year.

Patients who require a CVC for critical care in ICU will be recruited and randomly assigned to one of the two different groups to receive either a conventional non-impregnated CVC or an antimicrobial-impregnated CVC, which will be inserted and handled by medical practitioners. Participants will then be monitored for symptoms and signs of CLABSI, alongside length of ICU stay & healthcare costs. The diagnosis of CLABSI will be based on the CDC-NHSN (Centers for Disease Control and Prevention - National Healthcare Safety Network) definition. Researchers will then analyse and compare CLABSI rates and other relevant parameters among the 2 groups to see if antimicrobial-impregnated CVCs are useful and cost-effective in CLABSI prevention. Descriptive statistics will be expressed as percentages unless otherwise stated. Categorical variables will be expressed as percentages and compared using the Chi-square or Fisher's exact test, whichever is appropriate. Variables with a univariate test value of less than 0.05 (p-value) will be included in a multivariate analysis using a logistic regression model. Odds ratios (OR) and 95% confidence intervals (CI) will be calculated to identify the risk factors associated with the development of CLABSI in patients. In all instances, a p-value of less than or equal to 0.05 will be considered significant.

Local data at ICU, UMMC reported the incidence of CLABSI per 1000 catheter days in the first 6 months of 2022, to be 12.18. Using SAS (Statistical Analysis Software)® for sample size calculation, in order to detect a clinically significant reduction of CLABSI by 30%, and assuming a two-sided type I error protection of 0.05 and a power of 0.80, the calculated required sample size is 50 patients. To incorporate a 10% drop out rate, the study therefore aims to recruit 55 patients in each arm, making up to a total sample size of 110.

All data & information obtained in this study will be kept and handled in a confidential manner, in accordance with applicable laws and/or regulations.

The study hopes to demonstrate that the usage of antimicrobial-impregnated CVCs among adult critically ill patient in the ICU can reduce CLABSIs and this will translate to reduced patients' length of stay and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old and above who are admitted to the ICU of UMMC during the study period
* Patients who require a CVC during ICU stay

Exclusion Criteria:

* Patients who refuse to participate in the study
* Patients with known hypersensitivity reaction to CVC materials
* Patients with pre-existing diagnosis of CLABSI upon admission to the ICU
* Patients with pre-existing bloodstream infection upon admission to the ICU
* Patients with a pre-existing CVC, where sterility during placement may be compromised (e.g. in an emergency situation)
* Patients with indwelling CVC less than 48 hours
* Patients who had poor compliance to catheter bundle care during CVC handling throughout the indwelling catheter period
* Patients who require > 1 CVC or other central venous access

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Central line-associated bloodstream infection (CLABSI) rate | Through study completion, tentatively up to 1 year
  CLABSI cases per 1000 catheter days

SECONDARY OUTCOMES:
ICU Length of stay of patients diagnosed with CLABSI | Through study completion, tentatively up to 1 year
  Days of ICU stay
Healthcare costs of patients diagnosed with CLABSI | Through study completion, tentatively up to 1 year
  Healthcare costs, expressed in Malaysian Ringgit (MYR)
Percentages of specific bacterial species isolated from patients diagnosed with CLABSI | Through study completion, tentatively up to 1 year
  Percentages of specific bacterial species isolated from patients diagnosed with CLABSI
  Examples:
  * Gram positive organisms: Coagulase negative Staphylococci (CONS), Enterococci, Staphylococcus aureus
  * Gram negative organisms: Klebsiella, Pseudomonas, Escherichia coli, Acinetobacter
Percentages of antimicrobial resistance pattern groups among bacterial species isolated from patients diagnosed with CLABSI | Through study completion, tentatively up to 1 year
  Percentages of antimicrobial resistance pattern groups among bacterial species isolated from patients diagnosed with CLABSI
  Examples:
  * Methicillin Resistant Staphylococcus aureus (MRSA)
  * Extended-spectrum beta-lactamase (ESBL) producing Enterobacterales
  * Carbapenam-resistant Enterobacterales (CRE)
  * Multidrug-resistant Organisms (MRO)
  * Vancomycin-resistant Enterobacterales (VRE)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Ming Tan, Principal Investigator — University of Malaya
Locations (1):
- Universiti of Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang H, Tong H, Liu H, Wang Y, Wang R, Gao H, Yu P, Lv Y, Chen S, Wang G, Liu M, Li Y, Yu K, Wang C. Effectiveness of antimicrobial-coated central venous catheters for preventing catheter-related blood-stream infections with the implementation of bundles: a systematic review and network meta-analysis. Ann Intensive Care. 2018 Jun 15;8(1):71. doi: 10.1186/s13613-018-0416-4. PMID 29904809
- [Result] Lai NM, Chaiyakunapruk N, Lai NA, O'Riordan E, Pau WS, Saint S. Catheter impregnation, coating or bonding for reducing central venous catheter-related infections in adults. Cochrane Database Syst Rev. 2016 Mar 16;3(3):CD007878. doi: 10.1002/14651858.CD007878.pub3. PMID 26982376
- [Result] Lorente L, Lecuona M, Jimenez A, Lorenzo L, Diosdado S, Marca L, Mora ML. Cost/benefit analysis of chlorhexidine-silver sulfadiazine-impregnated venous catheters for femoral access. Am J Infect Control. 2014 Oct;42(10):1130-2. doi: 10.1016/j.ajic.2014.06.027. PMID 25278411
- [Result] Lorente L, Lecuona M, Jimenez A, Cabrera J, Santacreu R, Lorenzo L, Raja L, Mora ML. Chlorhexidine-silver sulfadiazine-impregnated venous catheters are efficient even at subclavian sites without tracheostomy. Am J Infect Control. 2016 Dec 1;44(12):1526-1529. doi: 10.1016/j.ajic.2016.04.236. Epub 2016 Jul 1. PMID 27378009
- [Result] Lorente L, Lecuona M, Jimenez A, Santacreu R, Raja L, Gonzalez O, Mora ML. Chlorhexidine-silver sulfadiazine-impregnated venous catheters save costs. Am J Infect Control. 2014 Mar;42(3):321-4. doi: 10.1016/j.ajic.2013.09.022. PMID 24581021
- [Result] Rosenthal VD, Duszynska W, Ider BE, Gurskis V, Al-Ruzzieh MA, Myatra SN, Gupta D, Belkebir S, Upadhyay N, Zand F, Todi SK, Kharbanda M, Nair PK, Mishra S, Chaparro G, Mehta Y, Zala D, Janc J, Aguirre-Avalos G, Aguilar-De-Moros D, Hernandez-Chena BE, Gun E, Oztoprak-Cuvalci N, Yildizdas D, Abdelhalim MM, Ozturk-Deniz SS, Gan CS, Hung NV, Joudi H, Omar AA, Gikas A, El-Kholy AA, Barkat A, Koirala A, Cerero-Gudino A, Bouziri A, Gomez-Nieto K, Fisher D, Medeiros EA, Salgado-Yepez E, Horhat F, Agha HMM, Vimercati JC, Villanueva V, Jayatilleke K, Nguyet LTT, Raka L, Miranda-Novales MG, Petrov MM, Apisarnthanarak A, Tayyab N, Elahi N, Mejia N, Morfin-Otero R, Al-Khawaja S, Anguseva T, Gupta U, Belskii VA, Mat WRW, Chapeta-Parada EG, Guanche-Garcell H, Barahona-Guzman N, Mathew A, Raja K, Pattnaik SK, Pandya N, Poojary AA, Chawla R, Mahfouz T, Kanj SS, Mioljevic V, Hlinkova S, Mrazova M, Al-Abdely HM, Guclu E, Ozgultekin A, Baytas V, Tekin R, Yalcin AN, Erben N. International Nosocomial Infection Control Consortium (INICC) report, data summary of 45 countries for 2013-2018, Adult and Pediatric Units, Device-associated Module. Am J Infect Control. 2021 Oct;49(10):1267-1274. doi: 10.1016/j.ajic.2021.04.077. Epub 2021 Apr 24. PMID 33901588

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT05959018/Prot_SAP_003.pdf
  • Informed Consent Form (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT05959018/ICF_001.pdf